CLINICAL TRIAL: NCT06899529
Title: Immediate Postoperative Bevacizumab Administration in Proliferative Diabetic Retinopathy Patients Undergoing Vitrectomy
Acronym: Postop IVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Ophthalmic Surgery Expedition Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IORG0009239-1
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Proliferative Diabetic Retinopathy - High Risk
Keywords: proliferative diabetic retinopathy; bevacizumab; vitreous hemorrhage
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Randomized Prospective Clinical Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and the specialist recording outcomes will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Active Comparator): Receives postoperative bevacizumab
  Interventions: Procedure: Bevacizumab
- Control Group (No Intervention): Does NOT receive postoperative bevacizumab

INTERVENTIONS:
Procedure: Bevacizumab — Bevacizumab will be given immediately after surgery in the Treatment Group
  Arms: Treatment Group

SUMMARY:
Patients undergoing surgery for complications related to diabetes will be recruited.

DETAILED DESCRIPTION:
Proliferative Diabetic Retinopathy patients undergoing pars plana vitrectomy will be randomized whether or not to receive intravitreal bevacizumab at the conclusion of the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is > 18
2. Subject consents to study participation and is capable of 6 months of follow-up.
3. The subject has type I or II Diabetes Mellitus with active PDR in the study eye.
4. Best-corrected spectacle visual acuity (BCSVA) on the Snellen eye chart ranges from 20/40 to Hand Motions in the study eye.
5. The subject is determined to need a PPV because of reduced BCSVA principally from a non-clearing vitreous hemorrhage, TRD, fibrous proliferation, or a combination of the three. When non-clearing vitreous hemorrhage is the principal reason for PPV, the hemorrhage must have been present by subjective history for at least 3 months. When TRD is the principal reason for PPV, the TRD must be threatening (within one disc diameter) or involving the fovea. When fibrovascular proliferation is the principal reason for PPV, it must be extensive (>3 clock hours) and threatening (within one disc diameter) or involving the fovea.
6. Only one eye per patient is eligible for the study.

Exclusion Criteria:

1. Subject is known to have a significant retinal/optic nerve disease otherwise unrelated to Diabetes Mellitus, which in the opinion of the examiner is responsible for two or more lines of reduced BCSVA (macular degeneration, optic neuritis, glaucoma, amblyopia, etc.) in the study eye.
2. Subject has a significant corneal opacity, which in the opinion of the examiner, is responsible for two or more lines of reduced BCSVA (corneal scar, ectasia, etc.) in the study eye.
3. Subject has had a previous vitrectomy (anterior or PPV) in the study eye.
4. Subject has uncontrolled neovascular glaucoma (intraocular pressure > 30 mmHg despite medical/surgical treatment) in the study eye.
5. Subject has uncontrolled hypertension (systolic > 200 mmHg or diastolic > 120 mmHg) despite adherence to a multiple anti-hypertensive medication regimen.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 6 months
  Postoperative vitreous hemorrhage rate

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Aleman, MD, Principal Investigator — Christian Ophthalmic Surgery Expedition Network
Locations (1):
- Sky Vision, Querétaro City, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Not sure at this point.

REFERENCES:
- [Background] Aleman I, Castillo Velazquez J, Rush SW, Rush RB. Ziv-aflibercept versus bevacizumab administration prior to diabetic vitrectomy: a randomised and controlled trial. Br J Ophthalmol. 2019 Dec;103(12):1740-1746. doi: 10.1136/bjophthalmol-2018-313313. Epub 2019 Jan 31. PMID 30705040
- [Background] Castillo Velazquez J, Aleman I, Rush SW, Rush RB. Bevacizumab before Diabetic Vitrectomy: A Clinical Trial Assessing 3 Dosing Amounts. Ophthalmol Retina. 2018 Oct;2(10):1010-1020. doi: 10.1016/j.oret.2018.04.014. Epub 2018 Oct 3. PMID 31047488
- [Background] Castillo J, Aleman I, Rush SW, Rush RB. Preoperative Bevacizumab Administration in Proliferative Diabetic Retinopathy Patients Undergoing Vitrectomy: A Randomized and Controlled Trial Comparing Interval Variation. Am J Ophthalmol. 2017 Nov;183:1-10. doi: 10.1016/j.ajo.2017.08.013. Epub 2017 Aug 30. PMID 28860046